CLINICAL TRIAL: NCT07241104
Title: A Phase I First-in-human Study to Investigate Safety, Tolerability, and Pharmacokinetics of AZD4063 in Adults With Phospholamban R14del Dilated Cardiomyopathy
Brief Title: A Study of AZD4063 in PLN R14del Dilated Cardiomyopathy
Acronym: PULSE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8340C00001
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Dilated Cardiomyopathy
Keywords: Single Ascending Dose; Multiple Ascending Dose; Phospholamban
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (SAD): Dose 1 of AZD4063 (Experimental): Participants will receive Dose 1 of AZD4063 via SC injection in Cohort 1 of SAD.
  Interventions: Drug: AZD4063
- Cohort 2 (SAD): Dose 2 of AZD4063 (Experimental): Participants will receive Dose 2 of AZD4063 via SC injection in Cohort 2 of SAD.
  Interventions: Drug: AZD4063
- Cohort 3 (SAD): Dose 3 of AZD4063 (Experimental): Participants will receive Dose 3 of AZD4063 via SC injection in Cohort 3 of SAD.
  Interventions: Drug: AZD4063
- Cohort 1 (MAD): Dose 4 of AZD4063 (Experimental): Participants will receive Dose 4 of AZD4063 via SC injection in Cohort 1 of MAD.
  Interventions: Drug: AZD4063
- Cohort 2 (MAD): Dose 5 of AZD4063 (Experimental): Participants will receive Dose 5 of AZD4063 via SC injection in Cohort 2 of MAD.
  Interventions: Drug: AZD4063
- Cohort 3 (MAD): Dose 6 of AZD4063 (Experimental): Participants will receive Dose 6 of AZD4063 via SC injection in Cohort 3 of MAD.
  Interventions: Drug: AZD4063
- Optional Cohort 1 (SAD): Dose 7 of AZD4063 (Experimental): Participants will receive Dose 7 of AZD4063 via SC injection in the optional cohort of the study. This additional cohort will be added depending on the findings.
  Interventions: Drug: AZD4063
- Optional Cohort 2 (SAD): Dose 8 of AZD4063 (Experimental): Participants will receive Dose 8 of AZD4063 via SC injection in the optional cohort of the study. This additional cohort will be added depending on the findings.
  Interventions: Drug: AZD4063
- Optional Cohort 1 (MAD): Dose 9 of AZD4063 (Experimental): Participants will receive Dose 9 of AZD4063 via SC injection in the optional cohort of the study. This additional cohort will be added depending on the findings.
  Interventions: Drug: AZD4063
- Optional Cohort 2 (MAD): Dose 10 of AZD4063 (Experimental): Participants will receive Dose 10 of AZD4063 via SC injection in the optional cohort of the study. This additional cohort will be added depending on the findings.
  Interventions: Drug: AZD4063

INTERVENTIONS:
Drug: AZD4063 — AZD4063 will be administered in the SAD and MAD part of the study as solution for injection via subcutaneous route of administration.

SUMMARY:
The purpose of the study is to assess the safety, tolerability and the pharmacokinetics (PK) of AZD4063 after single and multiple dose administration in participants with phospholamban (PLN) R14del dilated cardiomyopathy.

DETAILED DESCRIPTION:
This is a Phase 1, first in human, unblinded, ascending dose study which will be comprised of: 3 single ascending dose (SAD) cohorts, 3 multiple ascending dose (MAD) cohorts and optional cohorts.

The SAD part of the study will assess the single doses of AZD4063 across 3 cohorts. It will consist of:

* A screening period
* A treatment period: The participants will receive a single dose of AZD4063 by subcutaneous (SC) injection
* A follow-up period

The MAD part of the study will initiate on receiving the data from SAD cohort with available safety, PK and pharmacodynamics (PD) data from all cohorts. This part of the study will consist of:

* A screening period
* A treatment period: The participants will receive multiple doses of AZD4063 by SC injection
* A follow-up period

Optional cohorts may be added based on emerging safety, PK and PD data of the SAD and MAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 80 years of age inclusive, at the time of Screening
* Participants with pre-existing positive screening for R14 del PLN mutation
* Participants with screening Left ventricular eject fraction ≤ 45% as assessed by echocardiography
* Participants with New York Heart Association (NYHA) function class I-III
* Participants on stable medical therapy for at least 6 weeks prior to Screening and during the Screening period, with no significant improvement in heart failure
* Participants with implantable cardioverter-defibrillator (ICD) or Cardiac resynchronization therapy device (CRT-D)
* Participants with Body mass index (BMI) within the range 18-35 kg/m2
* Females of childbearing potential must not be lactating, and if heterosexually active must agree to use an approved method of highly effective contraception
* All females must have a negative pregnancy test at the Screening Visit.

Exclusion Criteria:

* Participants with positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody
* Known to have tested positive for Human immunodeficiency virus (HIV)
* Any known genetic mutation associated with hereditary electrical or structural disease
* Congenital long QT syndrome
* QTcF < 350 ms
* Known Short QT syndrome (SQTS) or family history of SQTS
* Catecholaminergic polymorphic ventricular tachycardia (CPVT as calcium ion channelopathy) and recent hospitalization for heart failure or significant ventricular arrhythmia within 3 months
* Participants with sustained ventricular arrhythmia requiring treatment and considered clinically not stable by the Investigator
* History of subendocardial Late Gadolinium Enhancement (LGE) suggestive of previous myocardial infarction and/or significant coronary artery disease (50% > stenosis in one major epicardial coronary artery or need for previous percutaneous coronary intervention or coronary artery bypass grafting)
* Routinely scheduled outpatient intravenous infusions for heart failure
* Uncontrolled hypertension
* Significant primary valvular disease
* Congenital heart disease
* Left ventricular wall thickness of > 13 mm or with any relative with hypertrophic cardiomyopathy (HCM)
* Recent acute presentation of myocarditis
* Restrictive or peripartum cardiomyopathy; infiltrative disorders (sarcoidosis)
* Alcohol consumption in excess
* Any laboratory values with the following deviations:

  1. Alanine Transaminase >2 upper normal limit (ULN)
  2. Aspartate Transaminase >2 ULN
  3. Total bilirubin > 2 x ULN
  4. Estimated GFR < 30 mL/min/1.73 m2
  5. Hemoglobin <10g/dL
* Any vital sign values with the following deviations at Screening

  1. Systolic blood pressure > 160 mmHg
  2. Diastolic blood pressure > 100 mmHg
  3. Pulse rate > 100 beats per minute
* Toxin exposure, systemic disease known to cause Dilated Cardiomyopathy (DCM)
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity
* Any history of cardiotoxic drug exposure with documented cardiomyopathy
* Noncardiac condition that limits expected lifespan to less than 1 year
* Participation in another clinical study with a study intervention administered in the last 3 months
* Participants with a known hypersensitivity to AZD4063
* Participants who are part of a gene therapy trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Cohort 1 (SAD): From Day 1 to Day 109, Cohorts 2 and 3 (SAD) From Day 1 to Day 99; For Cohorts 1,2 and 3 (MAD): Day 1 to Day 155
  The safety and tolerability of AZD4063 following the SC administration of single and repeated doses in participants with PLN R14del dilated cardiomyopathy

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from 0 to infinity (AUCinf) | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The AUCinf of single and repeated dose of AZD4063 following SC administration will be evaluated.
Area under the plasma concentration-curve from 0 to the last quantifiable concentration (AUClast) | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The AUClast of single and repeated dose of AZD4063 following SC administration will be evaluated.
Maximum plasma drug concentration (Cmax) | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The Cmax of single and repeated dose of AZD4063 following SC administration will be evaluated.
Renal clearance (CLR) | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The CLR of the single and repeated dose of AZD4063 following SC administration will be evaluated.
Cumulative amount of analyte excreted (Ae) | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The Ae of single and repeated dose of AZD4063 following SC administration will be evaluated
Fraction of dose excreted unchanged in urine (Fe) | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The Fe of single and repeated dose of AZD4063 following SC administration will be evaluated
Change in endomyocardial biopsy PLN messenger ribonucleic acid (mRNA levels) from baseline to estimated peak knockdown and estimated return-to-baseline | Cohort 1 (SAD): Up to Day 95, Cohorts 2 and 3 (SAD): Up to Day 85; Cohorts 1,2,3 (MAD): Up to Day 141
  The effects of single and repeated doses of AZD4063 on knockdown of PLN mRNA will be evaluated.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Rotterdam
  - Research Site, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/